CLINICAL TRIAL: NCT04220073
Title: Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Tolerability, Safety, Immunogenicity and Pharmacokinetic Profile of Single Dose of JS005 (Recombinant Humanized Monoclonal Antibody Against IL-17A) Injection in Healthy Volunteers
Brief Title: Phase I Study of Comparing Single Dose JS005 (Recombinant Humanized Monoclonal Antibody Against IL-17A) With Placebo in Tolerability, Safety, Immunogenicity and Pharmacokinetic in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: JS005-001
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Tolerability, Safety, Immunogenicity and Pharmacokinetic of JS005

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS005 (Experimental)
  Interventions: Biological: JS005 (recombinant humanized monoclonal antibody against IL-17A)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: JS005 (recombinant humanized monoclonal antibody against IL-17A) — JS005
  Arms: JS005
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
JS005-001 is one randomized, double-blind, placebo-controlled study to evaluate the tolerability, safety, immunogenicity and pharmacokinetic profile of single dose of JS005 injection in healthy volunteers.

A total of 5 dose groups are set in the study, i.e., 15 mg, 60 mg, 150 mg, 300 mg and 600 mg, single dose will be given subcutaneously in abdomen.

A total of 40 subjects are planned to be enrolled, 8 subjects will be enrolled in each group. Each dose group will be given the study drug and placebo at a ratio of 3:1. Each subject can only receive one single dose at one dose level.

Sentinel method will be used for dose escalation, and one independent safety evaluation team (SET) will be set up. 2 subjects (one receiving study drug, the other receiving placebo) will be randomized preferably and followed up until 3 days after administration when the dose starts in each dose group, the remaining 6 subjects (5 receiving study drug, 1 receiving placebo) can continue to be randomized after confirmation with the sponsor, if no any dose-limiting event (DLE) is observed during that period. Only when all the subjects at present dose level complete the follow-up for at least 14 days after administration, and no dose-limiting event (DLE) is observed in any one subject, the next dose level can be initiated after confirmation with the independent safety evaluation team and the sponsor, otherwise they must be observed for the full term of follow-up (i.e., on Day 85). If DLE is observed throughout the observational period, it is confirmed that ≤2/6 subjects have DLE after administration of the study drug through unblinding by the independent safety evaluation team, the next dose level can be initiated; if >2/6 subjects have DLE, the dose escalation will be terminated. The previous dose before that dose will be regarded as the maximum tolerated dose (MTD). When the dose for single dose is escalated to the preset maximum dose, and no safety endpoint is observed, it can be considered to continue to explore higher dose after joint decision by investigators and the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the informed consent form prior to the study, sufficient understanding of the content, course and possible adverse reactions of the study;
2. Being able to complete the study according to the requirements in the study protocol;
3. No plan of pregnancy and being willing to use effective contraceptive measures for subject (including partner) from 2 weeks prior to administration to 6 months after the last dose of study drug, see Appendix 5 for the specific contraceptive measures;
4. Male and female subjects aged 18 to 45 years, inclusive;
5. The body weight no less than 50 kg for male subjects and no less than 45 kg for female subjects. Body mass index (BMI) = weight (kg)/square of height, ranging from 18-26kg/m2 (including the critical value);
6. Normal or abnormal and clinically insignificant physical examination, vital signs;
7. Good health status, no history of cardiovascular, hepatic, renal, gastrointestinal, neurological, mental or metabolic disorders.

Exclusion Criteria:

1. Previous use of biopharmaceutical treatment directly targeting IL-17 monoclonal antibody or of IL-17 receptor (e.g., Secukinumab or Ixekizumab) at any time;
2. Use of therapeutic biological preparations within 12 weeks prior to administration (on Day 1), or remaining in the elimination period of the drug (within 5 half-lives) at randomization;
3. Participation in any other clinical study with intervention of investigational product within 12 weeks prior to randomization (on Day 1), or remaining in the elimination period of the drug (within 5 half-lives) at randomization;
4. Vaccination of Bacille Calmette-Guérin vaccine within 12 months prior to administration (on Day 1), or vaccination of other live vaccine within 12 weeks, or plan to use Bacille Calmette-Guérin vaccine or other live vaccine during the study and within 12 weeks after the study;
5. Any infection requiring hospitalization, antiviral or antibiotic therapy (e.g., pneumonia, cellulitis, bone and joint infection, etc., the subject is judged by investigators to have weakened immune system and may have unacceptable risk if participating in this study) within 30 days prior to administration (on Day 1);
6. Oral administration of herbal medicine within 30 days (inclusive), any prescription drug or over-the-counter drug, including Chinese herbal medicine for external use, vitamins and dietary supplements within 14 days (inclusive) prior to administration;
7. Any major surgery within 8 weeks (inclusive) prior to administration, or requiring such surgery during the study, and such surgery is considered by investigators to possibly bring unacceptable risk for subjects after confirmation by the sponsor;
8. Total white blood cell (WBC) count <3500/μl, platelet <100,000/μl, neutrophil <1500/μl or hemoglobin <8.5g/dL at screening;
9. Other clinically significant abnormality in clinical laboratory examination, or other clinical findings showing the following disorders of clinical relevance: including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immune, mental or cerebro- and cardiovascular diseases;
10. Abnormal ECG at screening (e.g., single QTc [QTcF]> 470 msec for male and > 480 msec for female) and/or other abnormalities of clinical significance, unacceptable risk that may be brought by participation in the study;
11. History of HIV infection, and/or positive HIV antibody, positive hepatitis B surface antigen (HBsAg), positive hepatitis C (HCV) antibody, or positive Treponema pallidum serum specific antibody (TP-CIA) at screening;
12. History of tuberculosis (TB) infection, or chest X-ray showing TB infection at screening, or tuberculosis screening (T-Spot) showing latent tuberculosis infection;
13. History of transplantation of vital organs (e.g., heart, lung, liver, kidney, etc.);
14. Having malignant tumors, not including the malignant tumors cured with no recurrence within the recent 5 years, completely resected basal cell and squamous cell carcinoma of skin, completely resected carcinoma in situ of any type);
15. Other major diseases within one year;
16. Positive urine drug screening, or history of drug abuse or use of narcotics in the past 5 years;
17. Positive alcohol test or intake of any alcohol-containing product within 48 hours prior to use of study drug;
18. History of excessive drinking or intake of excessive alcohol in the past 6 months (14 units of alcohol per week: 1 unit = 285mL beer, or 25ml liquor, or 100ml wine);
19. Known serious allergic reaction or hypersensitive to food, inhaled and contact material as well as drugs, or allergic constitution (allergy to various drugs and food);
20. Known history of allergy or hypersensitivity to the study drug, other monoclonal antibody drugs and therapeutic protein preparations (fresh or frozen plasma, human serum albumin, cytokine, interleukin etc.).
21. Female subjects with positive serum HCG or who are currently lactating;
22. Loss or donation of blood >400mL in recent three months, or receiving blood transfusion; or plan to donate blood during the study;
23. Any other condition that the subject is considered by investigators as inappropriate to participate in the study, for example, potential compliance issue, inability to complete all the tests and evaluations according to the requirements in the protocol, or uncontrolled mental, neurological or psychological disorders, participation in the study is judged by investigators to be associated with uncontrollable risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The minimum and maximum age of potential participants eligible for the clinical study, provided in relevant units of time
Enrollment: 40 (Estimated)
Dates: Start 2020-01-05 (Estimated); Primary Completion 2020-09-21 (Estimated); Study Completion 2021-01-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Clinically Significant Events . | From baseline through 12 weeks.
  Clinically significant events were defined as abnormal laboratory values and/or adverse events that are related to treatment.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Time to Reach the Maximum Concentration After Drug Administration (Tmax) in JS005 group.
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Observed Maximum Serum Concentration Following Drug Administration (Cmax) in JS005 group.
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Area Under the Serum Concentration-time Cure From Time Zero to the Time of Last Quantifiable Concentration (AUClast) in JS005 group.
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Area Under the Serum Concentration-time Curve From Time Zero to (AUCinf) in JS005 group.
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Mean residence time (MRT) in JS005 group.
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Systemic Clearance From Serum Following Intravenous Administration (CL) in JS005 group.
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Terminal Elimination Half-life (T1/2) in JS005 group
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Apparent terminal elimination rate constant in JS005 group.
Pharmacokinetics (PK) of JS005. | From baseline through 12 weeks.
  Apparent volume of distribution (Vd) in JS005 group.
Percentage of Participants With Anti-JS005 Antibodies. | From baseline through 24 weeks.
  Percentage of participants with treatment-emergent positive anti-JS005 antibodies was summarized by treatment group. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-JS005 antibodies / number of evaluable participants * 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Luhe Hospital Capital Medical University, Beijing, Beijing Municipality, China